CLINICAL TRIAL: NCT02042729
Title: A Phase 1 Comparative Study of E2022 Current and New Patch Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E2022-J081-006
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: volunteer

ARMS (4):
- E2022- Tape Formulation (Experimental)
  Interventions: Drug: E2022- Current Formula Tape
- Matching Placebo E2022 (Placebo Comparator): Matching Placebo
  Interventions: Drug: E2022 Matching Placebo- Current Formula Tape
- E2022- New Formulation (Active Comparator)
  Interventions: Drug: E2022- New Formula Tape
- Placebo E2022- New Formulation (Placebo Comparator): Matching Placebo
  Interventions: Drug: E2022 Matching Placebo- New Formula Tape

INTERVENTIONS:
Drug: E2022- Current Formula Tape — Cohort I: E2022 current formula tape administered on a skin application site and evaluated for 10 days during the introductory skin patch test.
  Cohort II: E2022 current formula tape administered to skin application site and evaluated for 20 days.
  Arms: E2022- Tape Formulation
Drug: E2022- New Formula Tape — Cohort I: E2022 new formula tape administered on a skin application site and evaluated for 10 days during the introductory skin patch test.
  Cohort II: E2022 new formula tape administered to skin application site and evaluated for 20 days.
  Arms: E2022- New Formulation
Drug: E2022 Matching Placebo- Current Formula Tape
  Other Names: Cohort I: E2022 Matching Placebo current formula tape administered on a skin application site and evaluated for 10 days during the introductory skin patch test.
  Arms: Matching Placebo E2022
Drug: E2022 Matching Placebo- New Formula Tape
  Other Names: Cohort I: E2022 Matching Placebo new formula tape administered on a skin application site and evaluated for
  Arms: Placebo E2022- New Formulation

SUMMARY:
The purpose of this study is to investigate the safety and pharmacokinetics of new patch formulation (tape) of E2022 by conducting patch test.

ELIGIBILITY:
Inclusion criteria

1. Non-smoker or not smoking for 4 weeks or longer before study treatment
2. BMI at screening is greater than or equal to 18.5 kg/m2 or less than 25.0 kg/m2
3. With written informed consent
4. Given full explanation of this study and is willing to and able to comply with study requirements.

Exclusion criteria

(Cohort 1 and 2):

1. Have a disorder which affects the evaluation of study drug such as psychiatric, gastrointestinal, hepatic, renal, respiratory, endocrinological, hematological, neurological, or cardiovascular system, or congenital metabolic abnormality
2. Have a clinically significant abnormality or organ dysfunction
3. Have a history of allergy to drug or food requiring medical treatment or seasonal allergy at screening
4. Have a history or complication of contact dermatitis or atopic dermatitis
5. Have hairy back or have shaved within 4 weeks before study treatment
6. Have a skin disease (e.g., eczema, dermatitis, dyschromatosis), or skin damage (e.g., injury, scar, or sun burn) which may affect skin assessment
7. Have a history or suspected to have drug or alcohol dependence, or positive for urine drug screen at baseline or a day before screening
8. Have had caffeine-containing drink or food, or alcohol within 72 hours before study treatment
9. Have used liquid product (including cosmetics), or applied patch, tape, or bandage on the back within 4 weeks before study treatment
10. Had hard exercise at least 5 days a week or a 1-hour or longer hard exercise within 2 weeks before study treatment

(Only Cohort 2):

1. Meet QTc of greater than 450 milliseconds at screening or immediately before study treatment
2. Had nutrients, herb preparations (e.g. oriental medicine), other food or drink (e.g., grapefruit-containing juice) which may affect the activity of drug-metabolizing enzyme or transporter within 2 weeks before study treatment
3. Had St. John's Wort-containing preparation within 4 weeks before Period 1 application

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 10 days (Cohort I) and 40 days (Cohort II)
Frequency of Adverse Events | 10 days (Cohort I) and 40 days (Cohort II)

SECONDARY OUTCOMES:
Pharmacokinetic Parameter: Cmax | 40 days (Cohort II)
Pharmacokinetic Parameter: Tmax | 40 days (Cohort II)
Pharmacokinetic Parameter: AUC | 40 days (Cohort II)

CONTACTS AND LOCATIONS:
Overall Officials: Hidetaka Hiramatsu, Study Director — Eisai Co., Ltd.
Locations (1):
- Fukuoka, Fukuoka, Japan